CLINICAL TRIAL: NCT06930599
Title: Comparison of Pulmonary Vein Isolation With and Without Transitional Zone Modification in Atrial Fibrillation Patients Without Low-Voltage Areas
Brief Title: Circumferential Pulmonary Vein Isolation Plus Transition Zone Modification in Atrial Fibrillation Patients Without Low-Voltage Areas
Acronym: PVI-TZM-AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Minglong Chen, Dr., The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-SR-1134
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Pulmonary vein isolation; Transition Zone Modification; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Follow-up physicians are blinded to treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Comparator: PVI-alone arm (Active Comparator)
  Interventions: Procedure: Pulmonary vein isolation alone
- Experimental: PVI+TZM arm (Experimental)
  Interventions: Procedure: Pulmonary vein isolation plus transition zone modification

INTERVENTIONS:
Procedure: Pulmonary vein isolation plus transition zone modification — For those who are randomized to PVI+TZM arm, additional TZM should be performed after finishing PVI ablation. PVI could be performed using open-irrigated contact-force catheter.
  Arms: Experimental: PVI+TZM arm
Procedure: Pulmonary vein isolation alone — In periprocedural period, all antiarrhythmic drugs were discontinued for at least 5 half-lives and amiodarone for 2 months before the procedure. An electrophysiological study was performed after overnight fasting and mild sedated state with administration of intravenous midazolam and fentanyl. PVI should be performed under the CARTO or Ensite electroanatomic mapping system using an open-irrigated contact-force ablation catheter.
  Arms: Active Comparator: PVI-alone arm

SUMMARY:
This study investigates two treatments for atrial fibrillation (AF) patients without low-voltage-areas (LVAs). It aims to determine whether adding transition zone modification (TZM) to the pulmonary vein isolation (PVI) improves long-term outcomes compared to PVI alone.

ELIGIBILITY:
Inclusion Criteria:

Aged 18 to 80 years AF referring for ablation No prior history of AF Absence of low-voltage areas during substrate mapping Presence of transition zone during substrate mapping Sign informed consent

Exclusion Criteria:

Presence of left atrial thrombus Acute coronary syndrome, cardiac surgery, angioplasty, or cerebrovascular accident within three months prior to enrollment Previous cardiac transplantation, complex congenital heart disease, rheumatic heart disease Untreated hypothyroidism or hyperthyroidism Dialysis-dependent terminal renal failure Life expectancy <12 months due to non-cardiovascular causes. Any conditions that, in the opinion of the investigator, may render the patient unable to complete the study Female under pregnancy or breast-feeding Involved in other studies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-04-09 (Estimated); Primary Completion 2026-10-09 (Estimated); Study Completion 2026-10-09 (Estimated)

PRIMARY OUTCOMES:
Freedom From AF and/or ATs With or Without Antiarrhythmic Drugs (AADs) | at least 12 months follow up
  Freedom from AF and/or ATs with or without antiarrhythmic drugs (AADs) at 12months after a single-ablation procedure. AF and/or AT occurring in the first 3 months after the ablation (blanking period) was censored. Each episode lasts > 30 seconds.

SECONDARY OUTCOMES:
Incidence of Peri-procedural Complications | 1 week after patient enrollment
  Incidence of Peri-procedural Complications：stroke, cardiac perforation, PV stenosis, esophageal injury and death
Total procedure time | 1 week after patient enrollment
  time that the patient spend in the procedure room
Total fluoroscopic time | 1 week after patient enrollment
  the total fluoroscopy time, during PVI alone or PVI plus low-voltage substrate modification
Total RF delivery time | 1 week after patient enrollment
  The cumulative duration (in minutes) of active radiofrequency (RF) energy application to the atrial tissue during the ablation procedure.

IPD SHARING:
Plan to Share IPD: Undecided